CLINICAL TRIAL: NCT00426673
Title: A Multi-Center, Open-Label, Unilateral Interaction Study of Ucb 34714 on Stable Phenytoin Monotherapy During a 45 Day b.i.d. Administration Period in 15 Adult Subjects Suffering From Epilepsy
Brief Title: An Open-Label Interaction Study to Look at the Effects of Brivaracetam on Phenytoin When Taken Together in 15 Adult Patients With Epilepsy.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01172
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-03

CONDITIONS: Epilepsy
Keywords: partial onset seizures, phenytoin, dilatin, brivaracetam, interaction
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

INTERVENTIONS:
Drug: Brivaracetam (ucb34714)

SUMMARY:
The primary objective of this Phase I study in 15 adult subjects suffering from epilepsy and chronically treated with phenytoin monotherapy is to evaluate the effect of steady-state ucb 34714 administration on the steady-state plasma levels of phenytoin.

ELIGIBILITY:
Inclusion Criteria:

* Well-characterized epileptic syndrome according to the ILAE classification.
* Patients currently treated with stable phenytoin monotherapy for at least three months and with at least one plasma measurement of pheyntoin within the target range (7 - 23 µg/ml) during the screening period.

Exclusion Criteria:

* History of status epilepticus in the last year.
* Subjects taking any drug that may significantly influence the metabolism of ucb 34714 (CYP2C or CYP3A potent inducers/inhibitors) except if the dose has been stable at least three months before entry into the study and will be kept stable for the entire trial duration.
* Subjects with a creatinine clearance of ≤50 mL/min.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
to evaluate the effect of steady-state ucb 34714 administration on the steady-state plasma levels of phenytoin.
Blood samples for PK calculations collected at different time points, on Visit 2 and Visit 7, for determination of phenytoin plasma concentrations (Phenytoin levels at pre-dose, 1, 2, 4, 6, 8, 12 (24 if PHT od) hours at V2 and V7)
The drug interaction on phenytoin will be assessed by comparison of AUCτ and Cmax between Visit 2 (phenytoin alone) and Visit 7 (combination of ucb 34714 and phenytoin).

SECONDARY OUTCOMES:
information on the tolerability and safety of the simultaneous administration of ucb 34714 and phenytoin in epilepsy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp von Rosenstiel, M.D., Study Director — UCB Pharma
Locations (3):
- United States (3):
  - Little Rock, Arkansas
  - Charlottesville, Virginia
  - Madison, Wisconsin